CLINICAL TRIAL: NCT00826735
Title: The Effect of Guided Imagery on the Third Stage of Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: Sigma Theta Tau International, Iota chapter (Unknown); Sigma Theta Tau International, Delta Psi chapter (Unknown); American College of Nurse-Midwive - ACNM Foundation (Industry)
Responsible Party: Mavis N. Schorn RN, CNM, PhD, Vanderbilt University School of Nursing
Purpose: Prevention
Other Study IDs: 070035
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2009-01

CONDITIONS: Third Stage of Labor; Bleeding; Guided Imagery; Childbirth
Keywords: third stage of labor; bleeding; guided imagery; childbirth
MeSH Terms: conditions — Hemorrhage | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Guided imagery (Experimental): The experimental group received a relaxation focused guided imagery intervention to use through the remainder of pregnancy plus a physiologic guided imagery intervention during the third stage of labor. These interventions were scripted and prerecorded on CDs.
  Interventions: Behavioral: Guided imagery

INTERVENTIONS:
Behavioral: Guided imagery — A relaxation focused guided imagery intervention was used through the remainder of pregnancy plus a physiologic guided imagery intervention was used during the third stage of labor.

SUMMARY:
The purpose of this study was to evaluate the effect of guided imagery on the third stage of labor. Blood loss from hemorrhage during childbirth, most commonly due to uterine atony, is one of the leading causes of maternal mortality in the United States and the leading cause of maternal death worldwide. The hypothesis was that the use of physiologic guided imagery would reduce the amount of bleeding during the third stage of labor.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older but less than 35 years
* English as her primary language
* fetus in a cephalic presentation
* singleton pregnancy
* 36 to 38 estimated gestational weeks
* no contraindications to vaginal delivery
* maternal weight less than 200 pounds prior to pregnancy

Exclusion Criteria:

* more than four previous children
* a history of postpartum hemorrhage
* bleeding disorder
* seizure disorder
* polyhydramnios
* diabetes (including gestational)
* hypertension
* cardiac disease
* uterine fibroids
* anemia (hematocrit less than 30)
* intrauterine fetal demise or tobacco use

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Blood Loss

SECONDARY OUTCOMES:
Length of third stage of labor

CONTACTS AND LOCATIONS:
Overall Officials: Mavis N Schorn, PhD, Principal Investigator — Vanderbilt University School of Nursing
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States